CLINICAL TRIAL: NCT00359099
Title: Proposal for Retrospective Review of the Prevalence of Hepatitis C Infection in Adult Patients Who Underwent Congenital Heart Surgery Before Screening
Brief Title: Hepatitis C in Adults Who Underwent Congenital Heart Surgery Before Screening
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: 0762-2006
Record Dates: First submitted 2006-07-31; First posted 2006-08-01 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Congenital Heart Disease
Keywords: Hepatic Medicine; Surgery
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This is a retrospective chart review. We hypothesize that patients who have undergone congenital heart surgery, prior to screening of blood products have a significant risk of hepatitis C infection and all such patients would benefit from screening for hepatitis C.

DETAILED DESCRIPTION:
The Adult Congenital Clinic at Emory Hospital routinely screens all patients who have had congenital heart surgery prior to 1992 for hepatitis C antibodies. It is currently not the practice norm for all congenital heart patients to receive hepatitis screening unless they are at a specialized clinic that has implemented a system. The question of hepatitis C serology is particularly important for this population as many of these patients develop heart failure and may require heart transplantation and immunosuppression.

This is a retrospective analysis examining the prevalence of hepatitis C in the Adult Congenital Clinic at The Emory Clinic. The current practice is to screen all adult congenital heart disease patients for hepatitis C. All Emory clinic charts reviewed will be of patients who had congenital heart surgery. Only information on patients who had surgery prior to 1992 will be used for this study. We will review approximately 1000 charts for this study.

ELIGIBILITY:
Inclusion Criteria:

* patients seen at Emory Adult Congenital Clinic
* patients > 18 years of age
* underwent surgery for congenital heart disease prior to 1992

Exclusion Criteria:

* history of known hepatitis prior to congenital heart surgery
* history of intravenous drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 1980-01; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: William T Mahle, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States